CLINICAL TRIAL: NCT05207046
Title: Role of ACCESsory Muscles in Mechanically Ventilated Patients After Spinal Cord Injury and Trauma: a Physiological Study - The ACCESSIT Study
Brief Title: The ACCESSIT Study
Acronym: ACCESSIT
Status: Recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 21-226
Record Dates: First submitted 2021-12-17; First posted 2022-01-26 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Support
Keywords: Spinal cord injury; Trauma; Respiratory muscles; Mechanical ventilation; Acute respiratory failure; Diaphragm dysfunction
MeSH Terms: conditions — Spinal Cord Injuries; Wounds and Injuries | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with spinal cord injury: Patients treated with mechanical ventilation after a traumatic spine lesion with spinal cord injury
  Interventions: Other: Mechanical Ventilation
- Patients with NO spinal cord injury: Patients treated with mechanical ventilation after a traumatic spine lesion with NO spinal cord injury
  Interventions: Other: Mechanical Ventilation

INTERVENTIONS:
Other: Mechanical Ventilation — Patients will be assessed and measurements will be taken during controlled ventilation (most likely <72 hours of ICU admission), during partially assisted ventilation, and until spontaneous unassisted breathing is reached.

SUMMARY:
The study is designed to characterize and monitor the structure, degree of activation and function of the different respiratory muscles during mechanical ventilation after spine trauma and spinal cord injury.

DETAILED DESCRIPTION:
In patients with spinal cord injury, separation from mechanical ventilation is an essential aspect of the prognosis. Denervation of specific muscles, as a consequence of the injury, can generate a dysfunction of the involved muscles and/or a disruption of their coordination during breathing. Respiratory muscle dysfunction is strongly associated with failure of weaning from mechanical ventilation. However, the pattern of activation and coordination of the different respiratory muscles, as well as their evolution over time, have been poorly investigated in spinal cord injury, particularly during the acute phase in intensive care unit.

Assessing the structure, activity, and function of the respiratory muscles at different time points after the injury would help to better understand the natural course of respiration in these patients and the possible therapeutic approaches. In fact, depending on the activation/deactivation and residual function of the respiratory muscles, there might be potential for recovery and training, with the possibility of improving patients' clinical outcomes.

In this preliminary physiological study, the investigators aim to assess the feasibility of monitoring non-invasively the respiratory muscles in mechanically ventilated adult patients with traumatic spine lesion, with and without spinal cord injury. The investigators also aim to assess, monitor, and compare over time the structure, degree of activation, function, and coordination of the different respiratory muscles.

Because the diagnosis of spinal cord injury is not always made immediately in spine trauma patients, and because other factors related to chest or abdominal trauma could interfere with the respiratory pattern, the plan is to study and follow patients with spinal cord injury, using patients with traumatic spine lesion without spinal cord injury as controls.

ELIGIBILITY:
Inclusion Criteria:

* Presence of traumatic spine lesion (with and without spinal cord injury)
* Requiring invasive mechanical ventilation, via oro-tracheal or tracheostomy tube,
* 16 years of age or older
* Patient or substitute decision maker able to provide consent

Exclusion Criteria:

* Expected withdrawal of treatments within 24 hours of screening
* Chronic respiratory failure already treated with mechanical ventilation before the injury
* Documented pre-existing neuromuscular diseases

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All mechanically ventilated patients with traumatic spine lesion (with and without spinal cord injury) will be considered for inclusion as early as possible after ICU admission (within 72 hours of admission).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Thickness and thickening fraction of the accessory muscles and their evolution over time during mechanical ventilation after spinal cord injury and spine trauma. | Baseline measurements assessed ≤ 72 hours from admission and subsequent measurements assessed > 72 hours from intensive care unit admission, until spontaneous unassisted breathing is reached, up to 6 weeks from enrollment
  Patients with spinal cord injury will be compared to patients with spine trauma and no spinal cord injury, at baseline and at different time points. The evolution of the ultrasound thickness of the respiratory muscles will also be compared to the evolution of the thickness of the limb muscles (rectus femoris). Regarding the primary outcome, patients with spinal cord injury will be compared to patients with spinal trauma and no spinal cord injury at baseline and at different time points. The evolution of the ultrasound thickness of the respiratory muscles will also be compared to the evolution of the thickness of the limb muscles (rectus femoris).

SECONDARY OUTCOMES:
Timing of activation and coordination of the diaphragm and of the different accessory muscles will be assessed using surface electromyography and monitored over time, after spinal cord injury and spine trauma. | > 72 hours after intensive care unit admission up to 6 weeks from enrollment
Rib cage and abdomen displacement and their coordination will be recorded and monitored over time using respiratory inductive plethysmography, after spinal cord injury and spine trauma. | > 72 hours after intensive care unit admission up to 6 weeks from enrollment
  Measures to be assessed will be: phase angle, asynchronies and/or paradox of rib cage and abdomen, maximum compartmental amplitude/tidal volume ratio, rib cage/tidal volume ratio (relative contribution of the rib cage to the tidal volume).

CONTACTS AND LOCATIONS:
Locations (1):
- Unity Health Toronto - St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No